CLINICAL TRIAL: NCT05497115
Title: Testing a Scalable Model of Care to Improve Patients Access to Mental Health Services After Traumatic Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: George Washington University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth Ruggiero, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20901; 1R01HS028006-01A1 (AHRQ)
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma Resilience and Recovery Program (Experimental): TRRP is a stepped model of care that delivers education at the bedside about mental health recovery after traumatic injury as well as risk assessment and brief intervention for high-risk patients (Step 1), fosters symptom monitoring and continued education (Step 2), screens for PTSD and depression 30 days post-injury (Step 3), and provides a referral and warm handoff to mental health services if needed (Step 4)
  Interventions: Behavioral: Trauma Resilience and Recovery Program
- Enhanced Usual Care Condition (No Intervention): Patients in the EUC arm will be given education about mental health after traumatic injury, educational materials about mental health recovery, and local referral information to assist treatment-seeking patients in seeking care.

INTERVENTIONS:
Behavioral: Trauma Resilience and Recovery Program — The Trauma Resilience and Recovery Program is a stepped model of care that is designed to deliver education at the bedside about mental health recovery after traumatic injury as well as risk assessment and brief intervention for high-risk patients (Step 1), foster symptom self-monitoring and continued education (Step 2), screen for PTSD and depression 30 days post-injury (Step 3), and provide a referral and warm handoff to mental health services if needed (Step 4).
  Arms: Trauma Resilience and Recovery Program

SUMMARY:
The purpose of this study to learn about patients' experience with the Trauma Resilience and Recovery program (TRRP) and/or the enhanced care group.

DETAILED DESCRIPTION:
In 2015, our team launched the Trauma Resilience and Recovery Program (TRRP) at the Medical University of South Carolina's Level I trauma center. TRRP is a stepped model of care that is designed to deliver education at the bedside about mental health recovery after traumatic injury as well as risk assessment and brief intervention for high-risk patients (Step 1), foster symptom self-monitoring and continued education via our automated text messaging system (Step 2), screen for PTSD and depression by chatbot or telephone 30 days post-injury (Step 3), and provide a referral and warm handoff to mental health services if needed (Step 4). The purpose of the proposed study is to examine the clinical and functional impact of TRRP over a period of 12 months. We will conduct a randomized controlled trial (RCT) with one-year follow up of TRRP vs. enhanced usual care (EUC) with 350 patients at The George Washington University (GWU) hospital, which serves a diverse population of ~2000 trauma center patients per year (15% penetrating mechanism). Trained, supervised interviewers blind to study condition will assess clinical and functional outcomes 3-, 6-, and 12-months post-baseline (Aim 1). Qualitative interviews will be conducted with ≥ 30 patients from underrepresented minority groups (i.e., African American, Latinx) as well as ≥ 20 victims of violent trauma (penetrating mechanism) to identify opportunities to strengthen the model to meet the diverse needs of these patients (Aim 2). GWU does not currently have an embedded mental health program in place, which will enable us to explore implementation determinants systematically (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking patients ≥ 16 years old who are admitted to George Washington University hospital's trauma center and screen positive on the Injured Trauma Survivors Screen (which indicates risk for development of posttraumatic stress disorder and/or depression) will be included.

Exclusion Criteria:

* Patients who have a Glasgow Coma Scale score under 13 at hospital admission, moderate to severe cognitive impairment (as measured by the Montreal Cognitive Assessment), active psychosis, or injury that prevents verbal communication (e.g., serious head or spinal cord injury) or is self-inflicted will be excluded. Patients with positive substance use screens via GWU's SBIRT protocol (~7% of the patient population) will be assessed by the clinical team with reference to severity and recency of substance use problems. We have found at MUSC that a high percentage of patients with SBIRT- positive screens are nevertheless good candidates for TRRP (>85%), but patients with serious, active substance abuse problems are likely not good candidates for TRRP and therefore will be excluded and referred to a substance use treatment center.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline PTSD Checklist for DSM-5 8- item (PCL8-5) at 3-,6-, and 12-month | Baseline, 3-, 6-, and 12- months post-baseline
  The PTSD Checklist for DSM-5 (Weathers et al., 2013) is a self-report measure that assesses the extent to which participants are bothered by the DSM-5 PTSD symptoms. Each symptom is rated on a scale of 0 (not at all) to 4 (extremely). Total scores are obtained by summing the scores of all items. The 8-item adaptation includes assessment of intrusive thoughts, avoidance of external reminders, negative expectations of self/ world, easily startled, emotional cue reactivity, avoidance of thoughts/emotions, loss of interest, and difficulty concentrating. The PCL8-5 has strong psychometric properties and clinical utility data similar to that of the long version.

SECONDARY OUTCOMES:
Demographics | Baseline
  Patients will provide standard demographic information, such as race/ethnicity; sex; gender identity; immigration, insurance, marital, and socioeconomic status; language; educational attainment; and occupation
Injured Trauma Survivor Screen (ITSS) | Baseline
  Injured Trauma Survivor Screen (ITSS) is a 9-item measure used to assess risk for development of posttraumatic stress symptoms following injury. Items are rated yes=1 and no=0. If the sum of questions 1, 2, 3, 5, and 6 is equal to or greater than 2, the screen is positive for PTSD risk. If the sum of questions 3, 4, 7, 8, and 9 is equal or greater than 2, the screen is positive for depression risk.
Electronic Medical Record Data (EMR) | Baseline
  Data will be collected at baseline via the electronic medical record including patients' length of stay; injury severity scores; number of emergency department visits; and opioid, anti-anxiety and anti-depression medications prescribed.
The Kessler 6 (K6) | Baseline, 3-, 6-, and 12- months post-baseline
  The Kessler 6 (K6) is a screening scale for nonspecific distress to discriminate cases of severe mental illness. Items are rated on a 5-point Likert scale (0-4). Total scores range from 0-24 and are calculated as the sum of all item ratings, with a total score ≥ 5 indicating moderate levels of distress and scores ≥ 13 indicating severe mental illness. This measure has been shown to have strong psychometric properties.
Patient Health Questionnaire-9 (PHQ-9) | 3-, 6-, and 12-months post- baseline assessment
  The Patient Health Questionniare-9 (PHQ-9) assesses the presence and frequency of 9 core depressive symptoms. Items are rated on a 4-point Likert scale (0-3). Total scores range from 0-27 and are calculated as the sum of all item ratings, with a total score of ≥ 10 indicating clinical significance.
PROMIS Emotional and Instrumental Support | Baseline, 3-, 6-, and 12- months post-baseline
  The PROMIS Emotion and Instrumental Support measure assesses perceived feelings of being cared for and valued as a person; having confidant relationships and availability of assistance with material, cognitive, or task performance.
  * Calculate a summed score across all items. All item responses scored on a scale of 1-5 where Never = 1, Always = 5
  * 3. Score of a 50 is the average for US population, SD of 10
PROMIS Self-Efficacy | 3-, 6-, and 12-months post- baseline assessment
  The 8-item PROMIS Self-Efficacy scale is a measure of confidence in one's ability to deal effectively with a variety of stressful situations.
  * Calculate a summed score access all items. All item responses scored on a scale of 1-5 where Never=1, Always = 5
  * Score of a 50 is the average for US population, SD of 10.
PROMIS Global Health | 3, 6, and 12-months post- baseline assessment
  The 10-item PROMIS Global Health questionnaire measures one's overall evaluation of one's physical and mental health.
PROMIS Pain Intensity and Interference Scale | 3-, 6-, and 12-months post- baseline assessment
  The PROMIS Pain Intensity and Interference scale assesses patients' pain and the extent to which it affects enjoyment of various activities in the past 7 days.
  * Calculate a summed score access all items. All item responses scored on a scale of 1-5 where Never=1, Always = 5
  * Score of a 50 is the average for US population, SD of 10.
PROMIS Sleep Disturbance | 3, 6, and 12-months post- baseline assessment
  The 4-item PROMIS Sleep Disturbance scale assesses perceptions of sleep quality, sleep depth, and restoration associated with sleep.
  * Calculate a summed score access all items. All item responses scored on a scale of 1-5.
  * Score of a 50 is the average for US population, SD of 10.
National Health Interview Survey Barriers to Care | Baseline, 3-, 6-, and 12- months post-baseline
  This protocol includes 5 interviewer-administered questions from the National Health Interview Survey (NHIS) Barriers to Care designed to assess when medical care was last sought, usual place of care, frequency of getting medical care and reasons for not getting medical care.
National Health Interview Survey Healthcare Utilization | Baseline and 12- months post-baseline
  This protocol includes interviewer-administered questions from the National Health Interview Survey (NHIS) Healthcare Utilization designed to assess when medical care was last sought, usual place of care, frequency of getting medical care and reasons for not getting medical care.
NHIS Mental Health Care Module | Baseline, 3-,6-, and 12-month post baseline
  6 items is designed to assess when mental health care was last sough, usual place of care, frequency of getting mental health care and reasons for not getting mental health care.
NHIS Job Status | Baseline, 3-,6-,and 12-month post baseline
  Consistent with Zatzick and colleagues (2008) we will ask patients about post-injury occupational status.
CMH SDOH items | Baseline, 3-,6-,12-month post baseline
  The Centers for Medicare & Medicaid Services (CMS) Center for Medicare and Medicaid Innovation (CMMI) made the Accountable Health Communities (AHC) Health-Related Social Needs (HRSN) Screening Tool to use in the AHC Model.1 The test is to see if systematically finding and dealing with the health-related social needs of Medicare and Medicaid beneficiaries has any effect on their total health care costs and makes their health outcomes better.
  The Tool can help providers find out patients' needs in these 5 core domains that community services can help with: Housing instability, food insecurity, transportation problems, Utility help needs and interpersonal safety.
The California Health Interview Survey (CHIS) question | Baseline, 3-, 6-, and 12- months post-baseline
  The California Health Interview Survey (CHIS) question allows a binary measurement of perceived prejudice, stereotyping, and discrimination in clinical encounters and experience.
Stigma Scale for Receiving Psychological Help | 3-month post- baseline assessment
  The Stigma Scale for Receiving Psychological Help assesses individuals' perceptions of how stigmatizing it is to receive psychological treatment. The SSRPH consists of 5 questions rated on a 4-point Likert scale.
  Total Score Instructions: Total score of the 5 items. No Items are reverse scored.
Discrimination in Medical Settings | 3-month post baseline
  The 7-item Discrimination in Medical Settings will measure perceived discrimination.
Collective Efficacy (Neighborhood Environment) | 3-months post-baseline
  The Neighborhood Environment Scale measures perceived neighborhood context and provides an estimate of cumulative exposure to adversity in childhood.
National Adverse Childhood Experiences Questions | 3-months post-baseline
  The six-item standard measure from the U.S. Department of Agriculture Economic Research Service is a validated, well-established measure of the availability, accessibility, and affordability of nutritionally adequate food.
NIDA Quick Screen (items 2-4); alcohol, tobacco, prescription and illicit drug use | 3-, 6-, and 12-months post- baseline assessment
  The NIDA Quick Screen is a validated instrument designed to assist providers in screening adults for substance use. The screen simply inquires whether a participant has used drugs (mood-altering, illegal, or prescription for nonmedical reasons), alcohol, or tobacco products within the past year and how often these substances have been used.
AUDIT-C | 3-,6-,12-month post baseline
  The Alcohol Use Disorders Identification Test (AUDIT-C) is an alcohol screen that can help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence).
Acceptance of Treatment Referral and Initiation of Treatment | 3-, 6-, and 12-months post- baseline assessment
  Patients will be asked whether they considered seeking assistance for mental health needs and whether they actually sought help. These questions will be based on semi-structured interviews administered via our needs assessment that were adapted from epidemiologic interviews conducted by our team in the aftermath of the September 11, 2001 terrorist attacks and recent natural disasters. Follow-up questions will inquire about whether patients sought help from family members, friends, chaplains, mental health professionals, or other health care professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ruggiero, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- George Washington University Hospital, Washington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
First, we will analyze the qualitative and quantitative data from our interviews and randomized controlled trial and will share these data via The National Database for Clinical Trials Related to Mental Illness. We will prepare both brief and comprehensive reports for AHRQ as we have done in prior NIH studies. We also will disseminate reports of our findings via print copy to the MUSC and GWU Public Relations office and websites. Additionally, we will prepare manuscripts for submission to research journals, such as JAMA, JAMA Surgery, JAMA Psychiatry, Am J Psychiatry, J Trauma and Acute Care Surgery, J Am College of Surgeons, Am J Public Health, and other sources that ensure broad dissemination. Additionally, as we have done previously with other federally funded grants, we will seek to present our findings to AHRQ staff and at national and international conferences.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available Year 3 quarter 3 of the study
Access Criteria: REDCap data dictionaries can be distributed for reuse at multiple institutions. A library of data dictionaries is made available for standards-based data collection forms and validated instruments. The underlying database is hosted in a secure data center at MUSC, a secure environment for data systems and servers on campus, and includes redundancy, failover capability, backups and extensive security checks.
URL: http://redcap.musc.edu

REFERENCES:
- [Background] Espeleta HC, Witcraft SM, Raffa T, Kartiko S, Dawson D, Becerra G, Roisman H, Hughes-Halbert C, Mueller M, Powell E, Brock T, Sarani B, Ruggiero KJ. Hybrid 1 randomized controlled trial of an integrated stepped-care mental health intervention for traumatic injury patients. Contemp Clin Trials. 2024 Nov;146:107694. doi: 10.1016/j.cct.2024.107694. Epub 2024 Sep 17. PMID 39299544

DOCUMENTS (1):
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT05497115/ICF_001.pdf